CLINICAL TRIAL: NCT05425797
Title: Building on Existing Tools To Improve Chronic Disease Prevention and Screening in Primary Care Virtually: the Virtual BETTER Study
Brief Title: The Virtual BETTER Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Kris Aubrey-Bassler, Associate Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CIHRVirtualBETTER
Record Dates: First submitted 2022-05-12; First posted 2022-06-21 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Delivery Modality of BETTER Intervention
Keywords: chronic disease; lifestyle; screening; physical activity; diet
MeSH Terms: conditions — Chronic Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: We will study two experimental groups (telephone and video) compared to the control group of in-person BETTER intervention delivery. Mode of delivery will be randomized between patients. If it is not feasible yo offer all three (e.g. PP only has capacity to offer virtual appointments, study population lives greater than 30 minutes travel from PP location), a subset of the three will be offered.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-Person (Active Comparator): Standard Prevention Practitioner visit that will take place in-person
  Interventions: Other: In-Person Prevention Practitioner Visit
- Video (Experimental): Prevention Practitioner visit that will take place through video call
  Interventions: Other: Video-Call Prevention Practitioner Visit
- Phone (Experimental): Prevention Practitioner visit that will take place through phone call
  Interventions: Other: Phone Prevention Practitioner Visit

INTERVENTIONS:
Other: In-Person Prevention Practitioner Visit — BETTER Intervention visit with PP which will take place in-person at the PP's office.
  Arms: In-Person
Other: Video-Call Prevention Practitioner Visit — BETTER Intervention visit with PP which will take place virtually via a secure video system.
  Arms: Video
Other: Phone Prevention Practitioner Visit — BETTER Intervention visit with PP which will take place via telephone.
  Arms: Phone

SUMMARY:
The focus of this project is to examine how delivering virtual care impacts health behaviour change for patients with chronic illnesses compared to in-person visits using a chronic disease prevention and screening (CDPS) program called BETTER (Building on Existing Tools To ImprovE Chronic Disease PRevention and Screening in Primary Care).

DETAILED DESCRIPTION:
While the current pandemic has launched a likely irreversible transition towards increased utilization of virtual methods for delivery of healthcare, we have only a very superficial understanding of how this shift will affect health outcomes and equity of access to health services. Several randomized trials comparing virtual to in-person delivery of health services have been completed, but none have examined the effect of interventions to address health behaviours, arguably one of the most challenging issues in healthcare and one that is most sensitive to the therapeutic relationship and modifiers to that relationship such as the mode of communication. The focus of this project is to examine how delivering virtual care impacts health behaviour change for patients with chronic illnesses compared to in-person visits using a chronic disease prevention and screening (CDPS) program called BETTER (Building on Existing Tools To ImprovE Chronic Disease PRevention and Screening in Primary Care).

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 40-70
* Persons who are already booking a BETTER prevention visit.

Exclusion Criteria:

* Persons with the presence of a terminal illness
* Persons in active treatment (i.e., systemic and/or radiation therapy) for cancer.
* Persons who are unable to provide informed consent.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Readiness to Change (University of Rhode Island Change Assessment Scale: URICA) | Post-Visit (less than 1 week after visit)
  To compare readiness to implement lifestyle change after telephone, video, and in-person BETTER Prevention visits.
  Min Score: 4 Max Score: 20
  Higher scores indicate a higher readiness to change (better outcome)

SECONDARY OUTCOMES:
Satisfaction of Modalities (Client Satisfaction Questionnaire: CSQ-4) | Post-Visit (less than 1 week after visit)
  To assess satisfaction with the three different delivery modalities.
  Min Score: 4 Max Score: 16
  Higher scores indicate higher satisfaction (better outcome)
Acceptability | Enrollment (Pre-visit)
  To assess acceptability of the three different delivery modalities.
  Assessed through enrollment questionnaire which will ask which delivery method they agree to. (Not scored on scale)
Accessibility | Enrollment (Pre-visit)
  To assess accessibility of the three different delivery modalities.
  Assessed through enrollment questionnaire which will ask why they chose which delivery method they did. (Not scored on scale)

CONTACTS AND LOCATIONS:
Overall Officials: Kris Aubrey-Bassler, MD, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Health Sciences Centre, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grunfeld E, Levine MN, Julian JA, Coyle D, Szechtman B, Mirsky D, Verma S, Dent S, Sawka C, Pritchard KI, Ginsburg D, Wood M, Whelan T. Randomized trial of long-term follow-up for early-stage breast cancer: a comparison of family physician versus specialist care. J Clin Oncol. 2006 Feb 20;24(6):848-55. doi: 10.1200/JCO.2005.03.2235. Epub 2006 Jan 17. PMID 16418496
- [Background] Grunfeld E, Julian JA, Pond G, Maunsell E, Coyle D, Folkes A, Joy AA, Provencher L, Rayson D, Rheaume DE, Porter GA, Paszat LF, Pritchard KI, Robidoux A, Smith S, Sussman J, Dent S, Sisler J, Wiernikowski J, Levine MN. Evaluating survivorship care plans: results of a randomized, clinical trial of patients with breast cancer. J Clin Oncol. 2011 Dec 20;29(36):4755-62. doi: 10.1200/JCO.2011.36.8373. Epub 2011 Oct 31. PMID 22042959
- [Background] Boekhout AH, Maunsell E, Pond GR, Julian JA, Coyle D, Levine MN, Grunfeld E; FUPII Trial Investigators. A survivorship care plan for breast cancer survivors: extended results of a randomized clinical trial. J Cancer Surviv. 2015 Dec;9(4):683-91. doi: 10.1007/s11764-015-0443-1. Epub 2015 Apr 21. PMID 25896265
- [Background] Elmslie K. Against the Growing Burden of Disease. Ottawa, ON: Public Health Agency of Canada.
- [Background] Grunfeld E, Manca D, Moineddin R, Thorpe KE, Hoch JS, Campbell-Scherer D, Meaney C, Rogers J, Beca J, Krueger P, Mamdani M; BETTER Trial Investigators. Improving chronic disease prevention and screening in primary care: results of the BETTER pragmatic cluster randomized controlled trial. BMC Fam Pract. 2013 Nov 20;14:175. doi: 10.1186/1471-2296-14-175. PMID 24252125
- [Background] Yarnall KS, Pollak KI, Ostbye T, Krause KM, Michener JL. Primary care: is there enough time for prevention? Am J Public Health. 2003 Apr;93(4):635-41. doi: 10.2105/ajph.93.4.635. PMID 12660210
- [Background] Grol R. Successes and failures in the implementation of evidence-based guidelines for clinical practice. Med Care. 2001 Aug;39(8 Suppl 2):II46-54. doi: 10.1097/00005650-200108002-00003. PMID 11583121
- [Background] Campbell-Scherer D, Rogers J, Manca D, Lang-Robertson K, Bell S, Salvalaggio G, Greiver M, Korownyk C, Klein D, Carroll JC, Kahan M, Meuser J, Buchman S, Barrett RM, Grunfeld E. Guideline harmonization and implementation plan for the BETTER trial: Building on Existing Tools to Improve Chronic Disease Prevention and Screening in Family Practice. CMAJ Open. 2014 Jan 22;2(1):E1-E10. doi: 10.9778/cmajo.20130040. eCollection 2014 Jan. PMID 25077119
- [Background] Tobe SW, Stone JA, Brouwers M, Bhattacharyya O, Walker KM, Dawes M, Genest J Jr, Grover S, Gubitz G, Lau D, Pipe A, Selby P, Tremblay MS, Warburton DE, Ward R, Woo V, Leiter LA, Liu PP. Harmonization of guidelines for the prevention and treatment of cardiovascular disease: the C-CHANGE Initiative. CMAJ. 2011 Oct 18;183(15):E1135-50. doi: 10.1503/cmaj.101508. Epub 2011 Sep 12. No abstract available. PMID 21911548
- [Background] Mair F, Whitten P. Systematic review of studies of patient satisfaction with telemedicine. BMJ. 2000 Jun 3;320(7248):1517-20. doi: 10.1136/bmj.320.7248.1517. PMID 10834899
- [Background] Whitten P, Love B. Patient and provider satisfaction with the use of telemedicine: overview and rationale for cautious enthusiasm. J Postgrad Med. 2005 Oct-Dec;51(4):294-300. PMID 16388172
- [Background] Bully P, Sanchez A, Zabaleta-del-Olmo E, Pombo H, Grandes G. Evidence from interventions based on theoretical models for lifestyle modification (physical activity, diet, alcohol and tobacco use) in primary care settings: A systematic review. Prev Med. 2015 Jul;76 Suppl:S76-93. doi: 10.1016/j.ypmed.2014.12.020. Epub 2015 Jan 5. PMID 25572619
- [Background] Grunfeld E, Moineddin R, Gunraj N, Del Giudice ME, Hodgson DC, Kwon JS, Elit L. Cancer screening practices of cancer survivors: population-based, longitudinal study. Can Fam Physician. 2012 Sep;58(9):980-6. PMID 22972732
- [Background] Pronk NP, Peek CJ, Goldstein MG. Addressing multiple behavioral risk factors in primary care. A synthesis of current knowledge and stakeholder dialogue sessions. Am J Prev Med. 2004 Aug;27(2 Suppl):4-17. doi: 10.1016/j.amepre.2004.04.024. PMID 15275669
- [Background] Coburn C, Collingridge D. Primary care and cancer: integration is key. Lancet Oncol. 2015 Sep;16(12):1225. doi: 10.1016/S1470-2045(15)00323-X. No abstract available. PMID 26431861
- [Background] Kelleher SA, Winger JG, Dorfman CS, Ingle KK, Moskovich AA, Abernethy AP, Keefe FJ, Samsa GP, Kimmick GG, Somers TJ. A behavioral cancer pain intervention: A randomized noninferiority trial comparing in-person with videoconference delivery. Psychooncology. 2019 Aug;28(8):1671-1678. doi: 10.1002/pon.5141. Epub 2019 Jun 19. PMID 31162756
- [Background] Armstrong AW, Chambers CJ, Maverakis E, Cheng MY, Dunnick CA, Chren MM, Gelfand JM, Wong DJ, Gibbons BM, Gibbons CM, Torres J, Steel AC, Wang EA, Clark CM, Singh S, Kornmehl HA, Wilken R, Florek AG, Ford AR, Ma C, Ehsani-Chimeh N, Boddu S, Fujita M, Young PM, Rivas-Sanchez C, Cornejo BI, Serna LC, Carlson ER, Lane CJ. Effectiveness of Online vs In-Person Care for Adults With Psoriasis: A Randomized Clinical Trial. JAMA Netw Open. 2018 Oct 5;1(6):e183062. doi: 10.1001/jamanetworkopen.2018.3062. PMID 30646223
- [Background] Arnedt JT, Conroy DA, Mooney A, Furgal A, Sen A, Eisenberg D. Telemedicine versus face-to-face delivery of cognitive behavioral therapy for insomnia: a randomized controlled noninferiority trial. Sleep. 2021 Jan 21;44(1):zsaa136. doi: 10.1093/sleep/zsaa136. PMID 32658298
- [Background] Befort CA, VanWormer JJ, Desouza C, Ellerbeck EF, Gajewski B, Kimminau KS, Greiner KA, Perri MG, Brown AR, Pathak RD, Huang TT, Eiland L, Drincic A. Effect of Behavioral Therapy With In-Clinic or Telephone Group Visits vs In-Clinic Individual Visits on Weight Loss Among Patients With Obesity in Rural Clinical Practice: A Randomized Clinical Trial. JAMA. 2021 Jan 26;325(4):363-372. doi: 10.1001/jama.2020.25855. PMID 33496775
- [Background] Clark DO, Keith N, Weiner M, Xu H. Outcomes of an RCT of videoconference vs. in-person or in-clinic nutrition and exercise in midlife adults with obesity. Obes Sci Pract. 2019 Feb 8;5(2):111-119. doi: 10.1002/osp4.318. eCollection 2019 Apr. PMID 31019728
- [Background] Guille C, Simpson AN, Douglas E, Boyars L, Cristaldi K, McElligott J, Johnson D, Brady K. Treatment of Opioid Use Disorder in Pregnant Women via Telemedicine: A Nonrandomized Controlled Trial. JAMA Netw Open. 2020 Jan 3;3(1):e1920177. doi: 10.1001/jamanetworkopen.2019.20177. PMID 32003816
- [Background] Lerdal A, Moe B, Digre E, Harding T, Kristensen F, Grov EK, Bakken LN, Eklund ML, Ruud I, Rossi JS. Stages of Change--continuous measure (URICA-E2): psychometrics of a Norwegian version. J Adv Nurs. 2009 Jan;65(1):193-202. doi: 10.1111/j.1365-2648.2008.04842.x. Epub 2008 Nov 14. PMID 19032513
- [Background] Pietrabissa G, Sorgente A, Rossi A, Simpson S, Riva G, Manzoni GM, Prochaska JO, Prochaska JM, Cattivelli R, Castelnuovo G. Stages of change in obesity and weight management: factorial structure of the Italian version of the University of Rhode Island Change Assessment Scale. Eat Weight Disord. 2017 Jun;22(2):361-367. doi: 10.1007/s40519-016-0289-1. Epub 2016 May 10. PMID 27165047
- [Background] Donner A, Birkett N, Buck C. Randomization by cluster. Sample size requirements and analysis. Am J Epidemiol. 1981 Dec;114(6):906-14. doi: 10.1093/oxfordjournals.aje.a113261. No abstract available. PMID 7315838
- See also: link to pubmed abstract for this pmid 16418496 — https://www.ncbi.nlm.nih.gov/pubmed/16418496
- See also: link to pubmed abstract for this pmid 22042959 — https://www.ncbi.nlm.nih.gov/pubmed/22042959
- See also: link to pubmed abstract for this pmid 25896265 — https://www.ncbi.nlm.nih.gov/pubmed/25896265
- See also: link to pubmed abstract for this pmid 24252125 — https://www.ncbi.nlm.nih.gov/pubmed/24252125
- See also: link to pubmed abstract for this pmid 12660210 — https://www.ncbi.nlm.nih.gov/pubmed/12660210
- See also: link to pubmed abstract for this pmid 11583121 — https://www.ncbi.nlm.nih.gov/pubmed/11583121
- See also: link to pubmed abstract for this pmid 25077119 — https://www.ncbi.nlm.nih.gov/pubmed/25077119
- See also: link to pubmed abstract for this pmid 21911548 — https://www.ncbi.nlm.nih.gov/pubmed/21911548
- See also: link to pubmed abstract for this pmid 10834899 — https://www.ncbi.nlm.nih.gov/pubmed/10834899
- See also: link to pubmed abstract for this pmid 16388172 — https://www.ncbi.nlm.nih.gov/pubmed/16388172
- See also: link to pubmed abstract for this pmid 25572619 — https://www.ncbi.nlm.nih.gov/pubmed/25572619
- See also: link to pubmed abstract for this pmid 22972732 — https://www.ncbi.nlm.nih.gov/pubmed/22972732
- See also: link to pubmed abstract for this pmid 15275669 — https://www.ncbi.nlm.nih.gov/pubmed/15275669
- See also: link to pubmed abstract for this pmid 26431861 — https://www.ncbi.nlm.nih.gov/pubmed/26431861
- See also: link to pubmed abstract for this pmid 30646223 — https://www.ncbi.nlm.nih.gov/pubmed/30646223
- See also: link to pubmed abstract for this pmid 32658298 — https://www.ncbi.nlm.nih.gov/pubmed/32658298
- See also: link to pubmed abstract for this pmid 33496775 — https://www.ncbi.nlm.nih.gov/pubmed/33496775
- See also: link to pubmed abstract for this pmid 31019728 — https://www.ncbi.nlm.nih.gov/pubmed/31019728
- See also: link to pubmed abstract for this pmid 32003816 — https://www.ncbi.nlm.nih.gov/pubmed/32003816
- See also: link to pubmed abstract for this pmid 19032513 — https://www.ncbi.nlm.nih.gov/pubmed/19032513
- See also: link to pubmed abstract for this pmid 27165047 — https://www.ncbi.nlm.nih.gov/pubmed/27165047